CLINICAL TRIAL: NCT00533507
Title: Primary Vaccination Course in Children Receiving the Pneumococcal Vaccine GSK 1024850A, Infanrix Hexa and Rotarix
Brief Title: Primary Vaccination Study With a Pneumococcal Conjugate Vaccine in Healthy Children 6 to 8 Weeks of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 109861
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Results first posted 2009-07-24 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-10

CONDITIONS: Infections, Rotavirus
Keywords: Pneumococcal vaccine.; Pneumococcal disease; Safety; Immunogenicity; Primary vaccination
MeSH Terms: conditions — Rotavirus Infections; Pneumococcal Infections | interventions — PHiD-CV vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; RIX4414 vaccine

ARMS (1):
- Synflorix group (Experimental): Subjects receiving Synflorix co-administered with Infanrix™ hexa at 1.5, 3 and 6 months of age, and co-administered with Rotarix™ at 1.5 and 3 months of age.
  Interventions: Biological: Synflorix; Biological: Infanrix hexa; Biological: Rotarix

INTERVENTIONS:
Biological: Synflorix — Intramuscular injection, 3 doses.
  Other Names: Pneumococcal conjugate vaccine GSK1024850A
Biological: Infanrix hexa — Intramuscular injection, 3 doses.
  Other Names: DTPa-HBV-IPV/Hib
Biological: Rotarix — Oral, 2 doses.
  Other Names: HRV vaccine

SUMMARY:
The purpose of this study is to assess the immunogenicity in terms of antibody response and the safety/reactogenicity in terms of solicited and unsolicited symptoms and serious adverse events following primary vaccination of Taiwanese infants with pneumococcal conjugate vaccine GSK 1024850A co-administered with a diphtheria, tetanus, acellular pertussis (DTPa)-combined vaccine and rotavirus vaccine in children during the first 6 months of life.

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including 6-8 weeks of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s) or guardian(s) of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of the study vaccines, or planned use during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before each dose of vaccines and ending 7 days after dose 1 and dose 2 and one month after dose 3.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* A family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, rotavirus and/or Streptococcus pneumoniae; with the exception of vaccines where the first dose may be given within the first two weeks of life according to the national recommendations (e.g. Hepatitis B and Bacillus Calmette-Guérin (BCG)).
* History of, or intercurrent, diphtheria, tetanus, pertussis, polio, hepatitis B and Haemophilus influenzae type b disease.
* Gastroenteritis within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal (GI) tract, intussusception (IS) or other medical condition determined to be serious by the investigator.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2007-09-18; Primary Completion 2008-06-01 (Actual); Study Completion 2008-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lin TY, Lu CY, Chang LY, Chiu CH, Huang YC, Bock HL, Tang H, Francois N, Moreira M, Schuerman L, Huang LM. Immunogenicity and safety of 10-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHiD-CV) co-administered with routine childhood vaccines in Taiwan. J Formos Med Assoc. 2012 Sep;111(9):495-503. doi: 10.1016/j.jfma.2011.07.014. Epub 2012 Mar 18. PMID 23021506
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109861 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synflorix Group
Started | 230
Completed | 229
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Synflorix Group
Number analyzed (Participants) | 230
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 6.4 (0.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 115

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Anti-Protein D Antibodies
Description: Concentrations are given as geometric mean concentrations (GMC) and expressed in Enzyme-Linked Immuno Sorbent Assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix Group
Number analyzed (Participants) | 219
EL.U/mL | 2277.6 [2048.7 to 2532.1]

2. Primary Outcome: Concentration of Anti-Pneumococcal Antibodies
Description: Concentrations are given as geometric mean titers (GMC) and expressed in microgram per milliliter (µg/mL).
  The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix Group
Number analyzed (Participants) | 219
µg/mL
  Anti-1 | 2.92 [2.65 to 3.22]
  Anti-4 | 3.79 [3.42 to 4.19]
  Anti-5 | 4.50 [4.11 to 4.93]
  Anti-6B | 1.69 [1.47 to 1.94]
  Anti-7F | 4.07 [3.72 to 4.46]
  Anti-9V | 3.90 [3.51 to 4.32]
  Anti-14 | 5.69 [5.10 to 6.35]
  Anti-18C | 7.28 [6.43 to 8.25]
  Anti-19F | 8.04 [7.37 to 8.78]
  Anti-23F | 2.81 [2.44 to 3.22]

3. Secondary Outcome: Number of Subjects With Anti-Protein D Antibody Concentrations Above the Cut-Off Value
Description: Anti-protein D antibody cut-off value assessed was greater than or equal to 100 Enzyme-Linked Immuno Sorbent Assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: Before the first dose (pre) and one month after (post) the third dose
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 219
subjects
  Pre (N=217) | 38
  Post (N=219) | 218

4. Secondary Outcome: Number of Subjects With Vaccine Pneumococcal Serotype Antibody Concentrations Above the Cut-Off Value
Description: Anti-pneumococcal antibody cut-off value assessed was 0.05 microgram per milliliter (μg/mL).
  The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: Before the first dose (pre) and one month after (post) the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 219
subjects
  Anti-1 Pre (N=217) | 111
  Anti-1 Post (N=219) | 219
  Anti-4 Pre (N=217) | 85
  Anti-4 Post (N=219) | 219
  Anti-5 Pre (N=217) | 149
  Anti-5 Post (N=219) | 219
  Anti-6B Pre (N=217) | 107
  Anti-6B Post (N=219) | 215
  Anti-7F Pre (N=218) | 138
  Anti-7F Post (N=219) | 219
  Anti-9V Pre (N=218) | 123
  Anti-9V Post (N=219) | 219
  Anti-14 Pre (N=218) | 203
  Anti-14 Post (N=219) | 219
  Anti-18C Pre (N=219) | 153
  Anti-18C Post (N=219) | 219
  Anti-19F Pre (N=219) | 172
  Anti-19F Post (N=219) | 219
  Anti-23F Pre (N=219) | 91
  Anti-23F Post (N=219) | 216

5. Secondary Outcome: Number of Subjects With Cross-Reactive Pneumococcal Serotype Antibody Concentrations Above the Cut-Off Value
Description: Anti-pneumococcal antibody cut-off value assessed was 0.05 microgram per milliliter (µg/mL).
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 219
subjects
  Anti-6A (N=219) | 210
  Anti-19A (N=218) | 200

6. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes Above the Cut-Off Value
Description: Cut-off value for opsonophagocytic activity against pneumococcal antibody assessed was greater than or equal to 1:8 titer.
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 103
subjects
  Opsono-1 (N=102) | 98
  Opsono-4 (N=103) | 103
  Opsono-5 (N=102) | 101
  Opsono-6B (N=102) | 89
  Opsono-7F (N=103) | 103
  Opsono-9V (N=98) | 98
  Opsono-14 (N=102) | 101
  Opsono-18C (N=101) | 99
  Opsono-19F (N=103) | 101
  Opsono-23F (N=102) | 98

7. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Cross-Reactive Pneumococcal Serotypes Above the Cut-Off Value
Description: as for outcome 6
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 97
subjects
  Opsono-6A | 87
  Opsono-19A | 38

8. Secondary Outcome: Number of Subjects With Anti-Polyribosyl-Ribitol Phosphate Antibody Concentrations Above the Cut-Off Value
Description: Anti-polyribosyl-ribitol phosphate antibody cut-off value assessed was greater than or equal to 0.15 microgram per milliliter (μg/mL).
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 58
subjects | 58

9. Secondary Outcome: Number of Subjects With Anti-Diphteria and Anti-Tetanus Toxoids Antibody Concentrations Above the Cut-Off Value
Description: Anti-diphteria and anti-tetanus toxoids antibody cut-off values assessed were greater than or equal to 0.10 International Units per milliliter (IU/mL).
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 58
subjects
  Anti-diphteria toxoid | 58
  Anti-tetanus toxoid | 58

10. Secondary Outcome: Number of Subjects With Anti-Pertussis (PT), Anti-Filamentous Hemagglutinin (FHA) and Anti-Pertactin (PRN) Antibody Concentrations Above the Cut-Off Value
Description: Anti-PT, anti-FHA and anti-PRN cut-off values assessed were greater than or equal to 5 Enzyme-Linked Immuno Sorbent Assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 58
subjects
  Anti-PT (N=58) | 58
  Anti-FHA (N=58) | 58
  Anti-PRN (N=57) | 57

11. Secondary Outcome: Number of Subjects With Anti-Hepatitis B Surface Antigen (HBs) Antibody Concentrations Above the Cut-Off Value
Description: Anti-HBs antibody cut-off value assessed was greater than or equal to 10 milli-International Units per milliliter (mIU/mL).
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 32
subjects | 32

12. Secondary Outcome: Number of Subjects With Anti-Poliovirus 1, 2 and 3 Antibody Titers Above the Cut-Off Value
Description: Anti-poliovirus 1, 2 and 3 antibody cut-off value assessed was greater than or equal to 1:8 titer.
Time Frame: One month after the third dose
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 44
subjects
  Anti-poliovirus 1 | 44
  Anti-poliovirus 2 | 44
  Anti-poliovirus 3 | 44

13. Secondary Outcome: Number of Subjects With Anti-rotavirus Immunoglobulin A Antibody Concentrations Above the Cut-Off Value
Description: Anti-rotavirus IgA antibody cut-off value assessed was greater than or equal to 20 Units per milliliter (U/mL).
Time Frame: Four months after the administration of the second dose of Rotarix™ vaccine
Population: Analysis was performed on ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 51
subjects | 44

14. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include diarrhoea, drowsiness, fever, irritability, loss of appetite, and vomiting
Time Frame: During the 4-day (Day 0-3) period after each dose
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 230
subjects
  Pain | 146
  Redness | 144
  Swelling | 139
  Diarrhoea | 7
  Drowsiness | 190
  Fever | 153
  Irritability | 203
  Loss of appetite | 159
  Vomiting | 55

15. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Time Frame: During the 31-day (Day 0-30) period after each dose
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 230
subjects | 95

16. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Up to one month after the third dose
Measure: Number; unit: subjects
Arm/Group | Synflorix Group
Number analyzed (Participants) | 230
subjects | 15

ADVERSE EVENTS:
Arm/Group | Synflorix Group
Serious Adverse Events (participants affected / at risk) | 15
Other Adverse Events (participants affected / at risk) | 224/230
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Synflorix Group
Urinary tract infection (Infections and infestations) | 6/230
Bronchiolitis (Infections and infestations) | 4/230
Gastroenteritis (Infections and infestations) | 2/230
Pyrexia (General disorders) | 2/230
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1/230
Bronchopneumonia (Infections and infestations) | 1/230
Dehydration (Metabolism and nutrition disorders) | 1/230
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1/230
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1/230
Enterocolitis (Gastrointestinal disorders) | 1/230
Gastroenteritis bacterial (Infections and infestations) | 1/230
Kawasaki's disease (Infections and infestations) | 1/230
Meningitis aseptic (Infections and infestations) | 1/230
Upper respiratory tract infection (Infections and infestations) | 1/230
Vesicoureteric reflux (Renal and urinary disorders) | 1/230
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Group (N=230)
Upper respiratory tract infection (Infections and infestations) | 54
Pain (General disorders) | 146
Redness (General disorders) | 144
Swelling (General disorders) | 139
Drowsiness (General disorders) | 190
Fever (General disorders) | 153
Irritability (General disorders) | 203
Loss of appetite (General disorders) | 159
Vomiting (General disorders) | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.